CLINICAL TRIAL: NCT03285425
Title: Natural History Study of Batten's CLN6 Disease
Brief Title: Natural History of Neuronal Ceroid Lipofuscinosis, Batten's CLN6 Diseae
Acronym: Batten'sCLN6
Status: Active, not recruiting | Type: Observational
Sponsor: Emily de los Reyes (Other)
Responsible Party: Sponsor-Investigator, Emily de los Reyes, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB16-00554
Record Dates: First submitted 2017-01-19; First posted 2017-09-18 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Batten Disease; CLN6
Keywords: Batten's disease; Neuronal Ceroid Lipofuscinosis
MeSH Terms: conditions — Neuronal Ceroid-Lipofuscinoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Natural history — Parent interview

SUMMARY:
CLN6 is a rare, neurodegenerative disease that causes progressive loss of acquired skills with motor delay, visual loss, seizures and ataxia. The investigators propose a natural history study of this rare disorder since it is currently unknown. It is important to understand disease progression in CLN6 disease to be able to judge therapeutic efficacy as emerging therapies like gene therapy become available.

DETAILED DESCRIPTION:
Neuronal Ceroid Lipofuscinosis (NCL) is the most common childhood neurodegenerative disorder characterized by accumulation of autofluorescent waxy lipopigments in the brain and other tissues. The symptoms manifest as blindness, seizures, ataxia, myoclonus and loss of milestones or dementia. This group of disorders caused by an intracellular accumulation of lipopigment (ceroid lipofuscin) material leads to neuronal death and is the most prevalent class of childhood neurodegenerative disease.

There are 14 types of NCL with 13 genotypes. Most of these are autosomal recessive. Neuronal ceroid lipofuscinosis, type 6 usually present like a late infantile NCL (CLN2) but can also present at as a juvenile onset (Mole). The natural history is not well established and the presentation maybe variable. There are currently no published data on the disease progression of children with CLN6 disease

CLN6 is a rare, neurodegenerative disease that causes progressive loss of acquired skills with motor delay, visual loss, seizures and ataxia. The investigators propose a natural history study of this rare disorder since it is currently unknown. Although there are descriptions of the clinical spectrum, the natural history has not been well described. It is important to understand disease progression in CLN6 disease to be able to judge therapeutic efficacy for as emerging therapies like gene therapy become available. The investigators will identify children with a genotypic diagnosis of CLN6 who are consulting Nationwide Children's hospital. The investigators will also recruit patients through family conferences of Batten's disease Support and Research association. The investigators propose a retro prospective chart review and longitudinal phone follow-up of with diagnosis of CLN6 to understand the onset and progression of this disease.

CLN6 is a rare, neurodegenerative disease that causes progressive loss of acquired skills with motor delay, visual loss, seizures and ataxia. The investigators propose a natural history study of this rare disorder since it is currently unknown. Although there are descriptions of the clinical spectrum, the natural history has not been well described. It is important to understand disease progression in CLN6 disease to be able to judge therapeutic efficacy for as emerging therapies like gene therapy become available. The investigators will identify children with a genotypic diagnosis of CLN6 who are consulting Nationwide Children's hospital. Patients will also be recruited through family conferences of Batten's disease Support and Research association.

OBJECTIVES:

The primary objectives of this study include the following:

1. Assess the natural history of CLN6 by performing a prospective, longitudinal chart review and phone follow-up of patients who have a diagnosis of Batten's disease, with a specific genotype of CLN6.
2. To promote better understanding of this disease to compare therapeutic efficacy with emerging therapies

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of genotypic diagnosis of CLN6

Exclusion Criteria:

* Patients who do not have a genotypic diagnosis of CLN6

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Study population will consist of children or adolescents (minors).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Natural history of disease progression | Three years
  The investigators will assess historical data for the onset of seizures, blindness, dementia, and loss of motor skills; and will request any available MRIs and EEGs.

CONTACTS AND LOCATIONS:
Overall Officials: Emily de los Reyes, MD, Principal Investigator — Abigail Wexner Research Institute, Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schulz A, Kohlschutter A, Mink J, Simonati A, Williams R. NCL diseases - clinical perspectives. Biochim Biophys Acta. 2013 Nov;1832(11):1801-6. doi: 10.1016/j.bbadis.2013.04.008. Epub 2013 Apr 17. PMID 23602993
- [Background] Canafoglia L, Gilioli I, Invernizzi F, Sofia V, Fugnanesi V, Morbin M, Chiapparini L, Granata T, Binelli S, Scaioli V, Garavaglia B, Nardocci N, Berkovic SF, Franceschetti S. Electroclinical spectrum of the neuronal ceroid lipofuscinoses associated with CLN6 mutations. Neurology. 2015 Jul 28;85(4):316-24. doi: 10.1212/WNL.0000000000001784. Epub 2015 Jun 26. PMID 26115733
- [Background] Sharp JD, Wheeler RB, Parker KA, Gardiner RM, Williams RE, Mole SE. Spectrum of CLN6 mutations in variant late infantile neuronal ceroid lipofuscinosis. Hum Mutat. 2003 Jul;22(1):35-42. doi: 10.1002/humu.10227. PMID 12815591
- [Background] Gao H, Boustany RM, Espinola JA, Cotman SL, Srinidhi L, Antonellis KA, Gillis T, Qin X, Liu S, Donahue LR, Bronson RT, Faust JR, Stout D, Haines JL, Lerner TJ, MacDonald ME. Mutations in a novel CLN6-encoded transmembrane protein cause variant neuronal ceroid lipofuscinosis in man and mouse. Am J Hum Genet. 2002 Feb;70(2):324-35. doi: 10.1086/338190. Epub 2001 Dec 21. PMID 11791207